CLINICAL TRIAL: NCT03799250
Title: Common Clinical Indices-guided Bolus-based vs. Continuous Fluid Management A Prospective, Randomized Trial
Brief Title: Fluid Management in the Post Anesthesia Care Unit
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 824-18
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2018-12

CONDITIONS: Ringer's Lactate
MeSH Terms: interventions — Ringer's Lactate; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Goal Directed Hemodynamic Therapy (Experimental): The GDT (Goal Directed Therapy) group will not receive any maintenance fluid. Fluid boluses will be given according to the flowchart attached.
  Baseline MAP and HR will be measured in the pre-anesthetic clinic or if not available will be recorded according to community medical record.
  Measurements of hemodynamic variables including heart rate and automatic non-invasive blood pressure measurements as well pulse oximetry as routine procedures will be recorded and stored by Metavision system (iMDsoft company) at regular intervals, all according to standard clinical practice.
  Blood gases measurement will be performed upon admission and at discharge. Urine output will be measured and recorded every hour.
  Other laboratory exams will be taken based on the physician discretion unrelated to the participation in the study.
  Interventions: Drug: Ringer lactate
- Control Group (Active Comparator): The control group will receive standard care which includes fluid maintenance program as dictated by the operating room anesthesiologist and as needed boluses through the PACU (Post Anesthesia Care Unit) stay.
  Interventions: Other: standard care

INTERVENTIONS:
Drug: Ringer lactate — Comparison between fluid maintenance in PACU compared to a bolus based goal directed hemodynamic therapy in the PACU
  Arms: Goal Directed Hemodynamic Therapy
Other: standard care — standard care
  Arms: Control Group

SUMMARY:
Fluid therapy is a cornerstone in patient therapy perioperatively. Many studies have addressed the amount of fluid administered (restrictive vs liberal strategies). Other studies focused on the type of fluids (colloid vs crystalloids), and in the last twenty years a more common subject of research was- the correct evaluation of the dynamic fluid status of patients.Bolus driven fluid therapy has been investigated in many goal-directed hemodynamic therapy (GDHT) trials and has become a widely used approach in intraoperative fluid management.

While there are numerous studies on the intraoperative outcome of GDHT, research on the immediate postoperative outcome of GDHT therapy use is scarce.

In this study the investigators aim to evaluate the efficacy of bolus-based fluid management guided by common clinical parameters in postoperative period in post-anesthesia care unit.

In this randomized clinical trial all patients will be randomized to one of the following groups:

The control group will receive standard care which includes fluid maintenance program as dictated by the operating room anesthesiologist and as needed boluses through the PACU stay.

The GDT group will not receive any maintenance fluid. Fluid boluses will be given according to the flowchart attached.

Measurements of hemodynamic variables including heart rate and automatic non-invasive blood pressure measurements as well pulse oximetry as routine procedures will be recorded and stored by Metavision system (iMDsoft company) at regular intervals, all according to standard clinical practice.

Blood gases measurement will be performed upon admission and at discharge. Urine output will be measured and recorded every hour.

DETAILED DESCRIPTION:
Methods Prior to surgery the patient will be assessed in the pre-anesthesia clinic, study protocol will be explained, questions answered and informed consent form will be signed by one of the investigating physicians. In case of an urgent case with no pre-anesthetic clinic visit, the process will take place in the entrance to the surgery room. Following surgery, patients will be assessed for eligibility and randomized to one of the study arms.

The control group will receive standard care which includes fluid maintenance program as dictated by the operating room anesthesiologist and as needed boluses through the PACU stay.

Study Arm:

The GDT group will not receive any maintenance fluid. Fluid boluses will be given according to the flowchart attached.

Baseline MAP and HR will be measured in the pre-anesthetic clinic or if not available will be recorded according to community medical record.

Blood products will be administered according to departmental guidelines and clinician decision unrelated to participation in the study.

Patients will be extubated, either in the operating room or postoperatively, when they fulfilled standard clinical criteria (adequate protective reflexes, adequate oxygenation, and stable hemodynamics), according to clinical indication unrelated to the participation in the study.

Measurements of hemodynamic variables including heart rate and automatic non-invasive blood pressure measurements as well pulse oximetry as routine procedures will be recorded and stored by Metavision system (iMDsoft company) at regular intervals, all according to standard clinical practice.

Blood gases measurement will be performed upon admission and at discharge. Urine output will be measured and recorded every hour.

Other laboratory exams will be taken based on the physician discretion unrelated to the participation in the study.

Data Collection:

For each participating patient the following data will be collected and recorded:

1. Demographic data
2. Medical history including regular medications
3. Hemodynamic data including heart rate, automatic non-invasive blood pressure measurements, temperature as well pulse oximetry as routine procedures will be recorded and stored by Metavision system
4. Anesthetic data including anesthetic method, anesthetic drugs, total fluid intake, anesthetic complications.
5. Laboratory values
6. Length of stay in PACU
7. Length of stay in hospital
8. Post-operative pulmonary complications
9. Acute kidney injury

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing general surgery, vascular surgery or urological surgery and who are expected to stay in the PACU for more than 8 hours.
* Above 18 years old
* Not requiring dialysis treatment
* Not requiring advanced monitoring (arterial waveform analysis or cardiac output monitoring)
* Eligible for signing an informed consent prior to surgery

Exclusion Criteria:

* - Pregnancy
* Inability to obtain an informed consent
* Massive transfusion in OR (more than 5 blood products)
* Colloids infusion needed
* The requirement for greater than 0.1mcg/kg/min of noradrenaline at arrival to PACU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The rate of postoperative complications measured according to the European Perioperative Clinical Outcome definitions and Clavien-Dindo Classification in the week following the intervention | 1 week post surgery
  Postoperative complication rates according to the EPCO classification

SECONDARY OUTCOMES:
The total amount of fluid infused. | 1 week post operative
Length of stay in PACU | 8 hours after surgery
Length of stay in hospital | 1 month after surgery
Post-operative pulmonary complications | 1 week after surgery
Acute kidney injury | 1 week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nadav O Sheffy, MD, Principal Investigator — Rabin Medical Center; Leonid O Eidelman, MD, Study Chair — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cecconi M, Corredor C, Arulkumaran N, Abuella G, Ball J, Grounds RM, Hamilton M, Rhodes A. Clinical review: Goal-directed therapy-what is the evidence in surgical patients? The effect on different risk groups. Crit Care. 2013 Mar 5;17(2):209. doi: 10.1186/cc11823. PMID 23672779
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Early goal-directed therapy after major surgery reduces complications and duration of hospital stay. A randomised, controlled trial [ISRCTN38797445]. Crit Care. 2005;9(6):R687-93. doi: 10.1186/cc3887. Epub 2005 Nov 8. PMID 16356219
- [Background] Della Rocca G, Vetrugno L, Tripi G, Deana C, Barbariol F, Pompei L. Liberal or restricted fluid administration: are we ready for a proposal of a restricted intraoperative approach? BMC Anesthesiol. 2014 Aug 1;14:62. doi: 10.1186/1471-2253-14-62. eCollection 2014. PMID 25104915
- [Background] Malbouisson LMS, Silva JM Jr, Carmona MJC, Lopes MR, Assuncao MS, Valiatti JLDS, Simoes CM, Auler JOC Jr. A pragmatic multi-center trial of goal-directed fluid management based on pulse pressure variation monitoring during high-risk surgery. BMC Anesthesiol. 2017 May 30;17(1):70. doi: 10.1186/s12871-017-0356-9. PMID 28558654
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Hand WR, Stoll WD, McEvoy MD, McSwain JR, Sealy CD, Skoner JM, Hornig JD, Tennant PA, Wolf B, Day TA. Intraoperative goal-directed hemodynamic management in free tissue transfer for head and neck cancer. Head Neck. 2016 Apr;38 Suppl 1(Suppl 1):E1974-80. doi: 10.1002/hed.24362. Epub 2016 Feb 1. PMID 26829494
- [Background] Calvo-Vecino JM, Ripolles-Melchor J, Mythen MG, Casans-Frances R, Balik A, Artacho JP, Martinez-Hurtado E, Serrano Romero A, Fernandez Perez C, Asuero de Lis S; FEDORA Trial Investigators Group. Effect of goal-directed haemodynamic therapy on postoperative complications in low-moderate risk surgical patients: a multicentre randomised controlled trial (FEDORA trial). Br J Anaesth. 2018 Apr;120(4):734-744. doi: 10.1016/j.bja.2017.12.018. Epub 2018 Feb 3. PMID 29576114
- [Background] Myles PS, Bellomo R, Corcoran T, Forbes A, Peyton P, Story D, Christophi C, Leslie K, McGuinness S, Parke R, Serpell J, Chan MTV, Painter T, McCluskey S, Minto G, Wallace S; Australian and New Zealand College of Anaesthetists Clinical Trials Network and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus Liberal Fluid Therapy for Major Abdominal Surgery. N Engl J Med. 2018 Jun 14;378(24):2263-2274. doi: 10.1056/NEJMoa1801601. Epub 2018 May 9. PMID 29742967
- [Background] Sanders GM. Randomized clinical trial assessing the effect of Doppler-optimized fluid management on outcome after elective colorectal resection (Br J Surg) 2006; 93; 1069-1076. Br J Surg. 2006 Dec;93(12):1563. doi: 10.1002/bjs.5683. No abstract available. PMID 17115398
- [Background] Weinberg L, Ianno D, Churilov L, Chao I, Scurrah N, Rachbuch C, Banting J, Muralidharan V, Story D, Bellomo R, Christophi C, Nikfarjam M. Restrictive intraoperative fluid optimisation algorithm improves outcomes in patients undergoing pancreaticoduodenectomy: A prospective multicentre randomized controlled trial. PLoS One. 2017 Sep 7;12(9):e0183313. doi: 10.1371/journal.pone.0183313. eCollection 2017. PMID 28880931
- [Background] Challand C, Struthers R, Sneyd JR, Erasmus PD, Mellor N, Hosie KB, Minto G. Randomized controlled trial of intraoperative goal-directed fluid therapy in aerobically fit and unfit patients having major colorectal surgery. Br J Anaesth. 2012 Jan;108(1):53-62. doi: 10.1093/bja/aer273. Epub 2011 Aug 26. PMID 21873370
- [Background] Van der Linden PJ, Dierick A, Wilmin S, Bellens B, De Hert SG. A randomized controlled trial comparing an intraoperative goal-directed strategy with routine clinical practice in patients undergoing peripheral arterial surgery. Eur J Anaesthesiol. 2010 Sep;27(9):788-93. doi: 10.1097/EJA.0b013e32833cb2dd. PMID 20613538
- [Background] Valentine RJ, Duke ML, Inman MH, Grayburn PA, Hagino RT, Kakish HB, Clagett GP. Effectiveness of pulmonary artery catheters in aortic surgery: a randomized trial. J Vasc Surg. 1998 Feb;27(2):203-11; discussion 211-2. doi: 10.1016/s0741-5214(98)70351-9. PMID 9510275
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542